CLINICAL TRIAL: NCT06766396
Title: Predictors for Discontinuation of Post Placental Intrauterine Contraceptive Device (PPIUCD) at Two-year Point With Implications for Population Stabilization in Pakistan
Brief Title: Predictors of PPIUCD Discontinuation at Two Years: A Clinical Study in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Tayyiba Wasim, Professor Obstetrics & Gynaecology, Services Institute of Medical Sciences, Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB/2017/373/SIMS
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Postpartum Contraception; Reproductive Health; Family Planning
Keywords: Postpartum intrauterine contraceptive device; maternal Health; Population stabilization; contraception

STUDY DESIGN:
Intervention Model Description: This study uses a single-group assignment model where all eligible postpartum women who consent to participate receive the intervention of postpartum intrauterine contraceptive device (PPIUCD) insertion. The intervention is provided either immediately postpartum for vaginal deliveries using Kelly's forceps or during cesarean section before uterine closure. Participants are followed prospectively for up to 24 months to evaluate continuation rates, complications, and reasons for discontinuation of PPIUCD.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postpartum Intrauterine Contraceptive Device (PPIUCD) Insertion (Experimental): Participants in this arm will receive the intervention of a postpartum intrauterine contraceptive device (PPIUCD) insertion. The PPIUCD will be inserted immediately postpartum for vaginal deliveries using Kelly's forceps under aseptic conditions or during cesarean section prior to uterine incision closure. All insertions will be performed by trained healthcare professionals to ensure consistency. Participants will be followed prospectively for up to 24 months to assess continuation rates, complications, and satisfaction with the method.
  Interventions: Device: Postpartum Intrauterine Contraceptive Device (PPIUCD).

INTERVENTIONS:
Device: Postpartum Intrauterine Contraceptive Device (PPIUCD). — Participants in the intervention arm will receive a postpartum intrauterine contraceptive device (PPIUCD) immediately after delivery. For vaginal deliveries, the PPIUCD will be inserted manually using Kelly's forceps under aseptic conditions, while for cesarean deliveries, the device will be inserted before uterine incision closure. All insertions will be performed by trained healthcare professionals

SUMMARY:
This prospective cohort study evaluated the continuation rates, complications, and satisfaction associated with postpartum intrauterine contraceptive devices (PPIUCDs) as a long-acting reversible contraception (LARC) method. Conducted in the Department of Obstetrics and Gynecology at Services Hospital, Lahore, Pakistan, from November 2017 to December 31, 2022, the study enrolled pregnant women attending antenatal care. Counseling was conducted using the GATHER technique, and informed consent was obtained before insertion. PPIUCDs were inserted postpartum during vaginal or cesarean deliveries by trained healthcare professionals. Follow-ups at 3, 6, 12, and 24 months assessed continuation rates, complications, and reasons for discontinuation.

DETAILED DESCRIPTION:
This prospective cohort study was conducted in the Department of Obstetrics and Gynecology at Services Hospital, Lahore, Pakistan, from November 2017 to December 31, 2022, after receiving ethical approval from the Institutional Review Board (Ref No. IRB/2017/373/SIMS). The study aimed to evaluate the continuation rates, complications, and satisfaction associated with postpartum intrauterine contraceptive devices (PPIUCDs) as a method of long-acting reversible contraception (LARC). The Government of Punjab provided contraceptive supplies free of cost to support the study.

Pregnant women attending antenatal care were recruited for the study after being educated about the importance of contraception using the GATHER counseling technique. Women who expressed interest in LARC, including PPIUCD, were provided detailed information about its benefits and risks. Informed consent was obtained, and their socio-demographic data were documented using a structured questionnaire. Willingness to participate was noted by stamping the antenatal cards of consenting women.

PPIUCDs were inserted immediately postpartum for both vaginal and cesarean deliveries. For vaginal deliveries, Kelly's forceps were used under aseptic conditions. During cesarean deliveries, PPIUCDs were inserted before the uterine incision was closed. All insertions were performed by healthcare providers trained by master trainers to ensure standardized techniques and minimize complications. Each participant received a follow-up card containing information about potential issues, such as irregular bleeding or difficulty in feeling the thread, and instructions to report these problems promptly.

The structured questionnaire developed for the study captured key socio-demographic and clinical information, including age, parity, education, occupation, monthly income, family size, and access to smartphones or Wi-Fi. Data on prior contraceptive use, reasons for non-use (e.g., myths or religious beliefs), and motivations for choosing PPIUCD (e.g., convenience, family influence, or doctor counseling) were also collected.

Participants were followed up at 3 months, 6 months, 1 year, and 2 years after insertion, either through in-person visits or telephonic interviews. During these follow-ups, data on complications such as irregular or heavy menstrual bleeding, pelvic pain, vaginal discharge, or device expulsion were recorded. Women were asked about their satisfaction with PPIUCD use and whether they continued or discontinued the method. For those who reported issues, a speculum examination was offered to check the thread position and trim it if necessary. Detailed information about device removal or expulsion, including the timing and reasons, was also collected during follow-ups.

The primary outcome of the study was the continuation rate at 24 months, defined as the probability of women consistently using the PPIUCD during this period. Secondary outcomes included reasons for discontinuation, and complications experienced.

Data analysis was performed using SPSS version 23. Qualitative variables were expressed as proportions with 95% confidence intervals (CIs). Comparative analyses between groups were conducted using the Chi-square test or Fisher's Exact test, depending on the data characteristics. A p-value of ≤ 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending antenatal care at the Department of Obstetrics and Gynecology, Services Hospital Lahore.
* Willing to use postpartum intrauterine contraceptive device (PPIUCD) as a method of contraception.
* Provided informed consent for participation in the study.
* Delivered via vaginal delivery or cesarean section with no contraindications to PPIUCD insertion.

Exclusion Criteria:

* Known uterine anomalies or severe uterine bleeding post-delivery.
* Diagnosed with chorioamnionitis or puerperal sepsis during delivery or postpartum.
* Known hypersensitivity or contraindications to copper-based intrauterine devices.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3400 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
continuation rate of PPIUCD at 24 months. | 24 months post-insertion
  The percentage of participants who continue using the postpartum intrauterine contraceptive device (PPIUCD) at 24 months after insertion.

SECONDARY OUTCOMES:
Complication Rate Associated with PPIUCD Use | From insertion to 24 months post-insertion
  The percentage of participants reporting complications such as heavy or irregular menstrual bleeding, expulsion, pelvic pain, or vaginal discharge during the follow-up period.
Reasons for PPIUCD Discontinuation | From insertion to 24 months post-insertion
  Documenting reasons for PPIUCD removal, including complications, misplaced ,wants another pregnancy or family pressures.
Expulsion Rate of PPIUCD | From insertion to 24 months post-insertion
  The percentage of participants experiencing spontaneous expulsion of the PPIUCD during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Tayyiba Wasim, FCPS, Principal Investigator — Services Institute of Medical Sciences, Pakistan
Locations (1):
- Services Institute of Medical sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No